CLINICAL TRIAL: NCT02950714
Title: Dissemination of the Lupus Interactive Navigator: Measuring Its Uptake and Impact on Global Health and Self-care
Brief Title: Dissemination of the Lupus Interactive Navigator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Paul Fortin, Professor of Medicine, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KAL-356634
Record Dates: First submitted 2016-10-19; First posted 2016-11-01 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIN_NOW (Experimental): Participants from CaNIOS centres randomized to the NOW group will be provided immediate access to the lupus interactive navigator (LIN), a web-based program developed to promote engagement and self-care in lupus.
  Interventions: Other: LIN_NOW
- LIN_WAIT (Active Comparator): Participants from CaNIOS centres randomized to the WAIT group will have usual care for three months prior to crossing over to access to the LIN.
  Interventions: Other: LIN_WAIT

INTERVENTIONS:
Other: LIN_NOW — The Lupus interactive navigator (LIN) was developed to facilitate and support engagement and self-management for persons with lupus. It is a web-based program that provides access to relevant information, resources, support, and other tools to help them manage their illness. It is accessible by the Internet and compatible for use with computer, tablet, and mobile device. The content for the LIN was based on the results of focus group discussions and web-based surveys of persons with lupus and health care providers. Medical researchers, writers, designers and programmers worked with clinical experts affiliated with the Canadian Network for improved outcomes in Systemic Lupus Erythematosus (CaNIOS) and persons with lupus to provide the written content and interview videos.
  Arms: LIN_NOW
Other: LIN_WAIT — Usual care for three months prior to access to the LIN
  Other Names: LIN at 3 months
  Arms: LIN_WAIT

SUMMARY:
This study asks whether persons with lupus will use and uptake the information and services of the web-based lupus interactive navigator (LIN) on a regular basis and whether this uptake will be associated with better self-management, improved coping, higher sense of control over their life, and overall improved health.

Systemic lupus erythematosus is an incurable chronic multi-organ inflammatory disease that affects preferentially young women. Unmet needs include a 15% excess in mortality, high morbidity and poor work outcomes. Despite prevalence of 1:2000, lupus is mostly unknown from the public and access to specialized care remains limited. Therefore, persons with lupus and their caregivers have difficulty finding high quality information relevant to their "lupus journey".

The LIN research team consists of a lupus clinical expert and researcher, a clinical psychologist and behavioral researcher, and a health information specialist. This team, funded by the Canadian Institutes of Health Research (CIHR), was responsible for the development of the LIN, a web-based navigator designed to promote self-care. The LIN is completed and the team will work with several stakeholders for dissemination: Lupus Canada, the Canadian Network for Improved Outcomes in Systemic Lupus Erythematosus (CaNIOS), the Arthritis Alliance of Canada, and lupus patient advisers. CaNIOS centres will be to randomized to immediate access to the LIN (LIN_NOW group) or usual care with crossover at 3 months (LIN_WAIT group). At baseline, all patients meeting entry criteria will be contacted, and asked to complete online questionnaires. At three months, a second online assessment will be performed before crossing over those from the centres randomized to usual care in order to now provide them with an access to the LIN. A final assessment will be performed at six months. Comparisons of baseline versus LIN exposure over three months will be performed in all patients at the end of the study; comparison of LIN use versus usual care will be done at three months; and retention of use at six months after LIN exposure will be documented in the first group randomized to LIN. The main outcome will be the Patient Activation Measure, a valid tool that measures the level of patient engagement. Secondary outcomes will include variables describing access and use of the LIN captured by the LIN server, coping, self-efficacy, and global health status.

DETAILED DESCRIPTION:
Self-management interventions are essential to meet the challenges of improving the care of persons with lupus and must be built on sound person-centered approaches aimed at self-empowerment. As such, patients need to be equipped with technology to provide them with relevant information and support tools. The Lupus Interactive Navigator (LIN) was developed to target these needs in persons with lupus. The LIN is a web-based program designed to provide relevant information and support engagement and self-management in lupus. The LIN was tested on 43 patients with lupus and yielded very high ratings for relevancy, credibility, and usefulness of the information provided and is now ready for dissemination.

An unblinded randomized cross-over study of the impact of the LIN will be performed. The study population will be restricted to patients enrolled in lupus clinics affiliated with the Canadian Network for Improved Outcomes in Systemic Lupus Erythematosus (CaNIOS). Centres will be randomized to be given access to the LIN at baseline (LIN_NOW) or be allocated to usual care with crossover to the LIN after a 3 month waiting period (LIN_WAIT) group. Following randomization, all participating CaNIOS centres will send a recruitment letter to all of their adult (18 years and older) lupus patients. The letter will explain that the nature of this national research project is aimed at measuring the usefulness of different support interventions in lupus.

Baseline: Patients willing to participate will be given instructions to access the survey website where they will be provided with consent and questionnaires to complete. following completion of the baseline questionnaires, patients in the LIN_NOW group will be given access to the LIN. Patients in the LIN_WAIT group will continue with usual care for three months.

Three months: Email reminders will be sent to all participants prior to the due date of the three month questionnaires. All email reminders will include the website link, instructions to access the user. The LIN-NOW group will continue with access to the LIN upon completion of these questionnaires. The LIN_WAIT group will continue with usual care for three months and cross over to the LIN upon completion of these questionnaires.

Six months: Email reminders will be sent to all participants to complete the third set of questionnaires prior to the due date.

Both NOW and WAIT groups will continue with access to the LIN upon completion of these questionnaires.

Measures: Questionnaires will include assessments of socio-demographic variables, patient activation, disease-related variables including self-reported disease activity and damage, coping, self-efficacy, mood and general health status. Four of the four main outcome measures relevant to this study will be, as follows:

The Patient Activation Measure PAM): The PAM is a 13-item that measures level of patient engagement in health care. This tool is designed to measure an individual's level of confidence, beliefs, knowledge, and skills about managing one's health. Respondents can answer with varying levels of agreement or disagreement on a 4-point Likert-type scale. This scale has been shown to have strong psychometric properties. The PAM has been used in observational and intervention studies as a patient-centered measure to monitor changes in patient's experiences over time, with higher scores related to greater self-management, healthy behaviors, medication adherence, better clinical outcomes and higher levels of satisfactions with services.

The Processes of Care Survey - Short Form (IPC-SF) assesses three domains of patient interpersonal centered care: communication, decision making, and interpersonal style. The following scales of the IPC-SF will be used: communication scales (lack of clarity, elicited concerns/responded, and explained results), patient-centered decision making scale, and one interpersonal style scale (compassionate/respectful). Higher scores indicate more reports of experiences of the specific dimension, such as more explanations or more instances of deciding together.

The Lupus Self-efficacy Scale (LSES) will measure patients' confidence related to lupus-specific domains. This 11-items version assesses level of confidence in managing or decreasing lupus-related symptoms (i.e. fatigue, mood). The construct and concurrent validity of this scale has been demonstrated . Self-efficacy has been found to be an important determinant in understanding the adoption of self-management approaches among patients with arthritis.

The Morisky Adherence Scale is a 4-item generic scale that may apply to all medications and diseases and does not measure any particular time frame.

Analysis. Descriptive statistics will be performed including a description of the use of LIN (number of visits, number of pages visited, number of minutes spent, etc). The first set of analyses will determine the impact of the LIN on the PAM, the primary outcome, for the entire population by comparing scores of both groups before and following a 3 month exposure to the LIN (differences in scores at 3 months versus baseline in LIN_NOW group pooled with the scores at 6 months versus 3 months in the LIN-WAIT group). Secondary analyses using the same predictor variable, the LIN, to determine the impact of the IPC-SF, LSES, and the Morisky scale, replacing the PAM as the outcome variable in those analyses. For each outcome variable, the analysis will compare mean differences in scores of the PAM at 3 months versus baseline. Multivariate analysis will control for demographic and clinical variables such as age, sex, education, access to internet, type of device use, disease duration, lupus activity, lupus damage, physical and mental health status, coping and social support. The second set of analyses will question whether there is a difference between exposure to the LIN and usual care by comparing the patients from the centres randomized to the use of the LIN in the first three months versus those from the centres randomized to usual care during that same period of time. The third sets of analyses will examine whether the impact that may be observed at three months in the group randomized to LIN now is sustained at six months by comparing the outcome measures at three and six months in the LIN_NOW group.

ELIGIBILITY:
Inclusion Criteria: Two levels of entry criteria are to be considered: 1) at the centre level and 2) at the patient level.

Centre level:

1. to have a centre affiliation with the Canadian Network for improving outcomes in Systemic Lupus Erythematosus (CaNIOS) and a lupus clinical expert who is an active member of CaNIOS willing to sign the letter of invitation,
2. to have a list of patients with contact information (mailing or an electronic address)
3. to have research staff available to prepare and submit this study to the local research ethics board.

Patient level:

1. ≥18 years of age
2. Diagnosis of Systemic Lupus Erythematosus (SLE) by the American College of Rheumatology (ACR) classification criteria, OR the new Systemic Lupus International Collaborating Clinics criteria (SLICC), OR deemed to have SLE by the treating physician
3. Able to read and write in English or French
4. Able to provide informed consent
5. Able to provide contact information (postal mail and email)
6. Able to complete online questionnaires.

Exclusion Criteria: Those that do not meet entry criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 541 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | Baseline, three and six months evaluations. Final evaluation at six months.
  The widely used 13-item PAM measures level of patient engagement in their healthcare [Development and testing of a short form of the patient activation measure. The tool is designed to measure an individual's level of confidence, beliefs, knowledge, and skills about managing one's health. Respondents can answer with varying levels of agreement or disagreement on a 4-point Likert-type scale. This scale has been shown to have strong psychometric properties. The PAM has been used in observational and interventional studies as a patient-centered measure to monitor changes in patient's experiences over time, with higher scores related to greater self-management, healthy behaviors, medication adherence, better clinical outcomes and higher levels of satisfactions with services. Between and within group changes in PAM scores over time of LIN exposure will be compared.

SECONDARY OUTCOMES:
Lupus self-efficacy scale (LSES) | Baseline, three and six months
  The LSES adapted for lupus from the Arthritis Self-efficacy Scales will measure patients' confidence related to lupus-specific domains. This 11-items version assesses level of confidence in managing or decreasing lupus-related symptoms (i.e. fatigue, mood). The construct and concurrent validity of this scale has been demonstrated. Self-efficacy has been found to be an important determinant in understanding the adoption of self-management approaches among patients with arthritis. Between and within group changes in LSES scores over LIN exposure will be compared.
Coping with Health Injuries and Problems (CHIP) | Baseline, three and six months
  This 32-item questionnaire assesses coping strategies typically used when coping with health problems. Its four sub-scales include distraction, palliative, instrumental coping, and emotional coping. This instrument has been shown to have good psychometric properties and has been recommended for use with different medical populations. Between and within group changes in CHIP scores over LIN exposure will be compared.
Health status measured by the SF-36 version 1 | Baseline, three and six months.
  This generic measure has been recommended for use in lupus, as it is both valid and reliable. It consists of a self-administered instrument with 36 questions that cover eight dimensions of well-being: physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. Besides scoring for each of the eight domains, an algorithm also allows calculation of normalized scores for physical and mental function, the physical component score (PCS) and the mental component score (MCS). Between and within group changes in SF-36 version 1 scores over LIN exposure will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Fortin, MD,MPH,FRCPC, Principal Investigator — CHU de Quebec-Universite Laval
Locations (10):
- Canada (10):
  - Calgary Health Sciences Centre, Calgary, Alberta
  - Edmonton University of Alberta, Edmonton, Alberta
  - Vancouver Arthritis Research Centre, Vancouver, British Columbia
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Hamilton McMaster University, Hamilton, Ontario
  - London St. Joseph Health Sciences Centre London, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre de recherche du CHU de Québec - université de Laval, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fortin PR, Neville C, Julien AS, Rahme E, Haroun V, Nimigon-Young J, Morrison AL, Eng D, Peschken CA, Vinet E, Hudson M, Smith D, Matsos M, Pope JE, Clarke AE, Keeling S, Avina-Zubieta JA, Rochon M, Da Costa D. Measuring the Impact of MyLupusGuide in Canada: Results of a Randomized Controlled Study. Arthritis Care Res (Hoboken). 2023 Mar;75(3):529-539. doi: 10.1002/acr.24871. Epub 2022 Nov 17. PMID 35225436